CLINICAL TRIAL: NCT04196387
Title: Antimicrobial Resistance Rate In Escherichia Coli And Klebsiella Pneumonia : A Retrospective Study
Status: Completed | Type: Observational
Sponsor: Batool Mutar (Other)
Responsible Party: Sponsor-Investigator, Batool Mutar, Prof Dr Batool Mutar Mahdi, Al-Kindy College of Medicine
Organization: Al-Kindy College of Medicine (Other)
Other Study IDs: 8 Al-KindyCM
Record Dates: First submitted 2019-12-07; First posted 2019-12-12 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Antibiotic Reaction
Keywords: antibiotics, urine, resistance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: urine culture — urine culture and antibiotic susceptibility test

SUMMARY:
Antibiotics are medicines used to avoid and treat bacterial infections. Antibiotic resistance is increasing to dangerous level globally.

DETAILED DESCRIPTION:
Antibiotics resistance is a global health problem.

ELIGIBILITY:
Inclusion Criteria:

1. patients with UTI
2. patients with dysuria
3. patients with loin pain

Exclusion Criteria:

1. patients with surgery
2. patients with cancer

Ages: 6 Months to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with dysurea
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
urine culture results | 3 years
  type of bacterial strain was isolated

IPD SHARING:
Plan to Share IPD: Undecided